CLINICAL TRIAL: NCT05599932
Title: A Phase 1, Open-label, Multi-center, Single-dose, Parallel Group Study to Evaluate the Pharmacokinetics of Siremadlin (HDM201) in Participants With Mild, Moderate and Severe Hepatic Impairment Compared to Matched Healthy Control Participants
Brief Title: Pharmacokinetics and Safety Study of Siremadlin (HDM201) in Participants With Mild, Moderate and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201X2105
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Solids tumors; Hematological malignancies; Child-Pugh classification; HDM201; Siremadlin
MeSH Terms: conditions — Hematologic Neoplasms | interventions — siremadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Healthy Control (Experimental): Each healthy participant will receive a single dose of HDM201
  Interventions: Drug: Siremadlin
- Group 2: Mild; Child-Pugh A (Experimental): Each participant with mild Child-Pugh will receive a single dose of HDM201
  Interventions: Drug: Siremadlin
- Group 3: Moderate; Child-Pugh B (Experimental): Each participant with moderate Child-Pugh will receive a single dose of HDM201
  Interventions: Drug: Siremadlin
- Group 4: Severe; Child-Pugh C (Experimental): Each participant with severe Child-Pugh will receive a single dose of HDM201
  Interventions: Drug: Siremadlin

INTERVENTIONS:
Drug: Siremadlin — HDM201 capsule
  Other Names: HDM201

SUMMARY:
The main purpose of this study is to evaluate the effect of varying degrees of impaired hepatic function (by Child Pugh classification) on the plasma PK of siremadlin after a single oral dose. In addition, safety and tolerability of siremadlin after a single oral dose will be evaluated. The results of this study will inform the decision whether a dose adjustment may be recommended when treating patients with various degrees of impaired hepatic function.

DETAILED DESCRIPTION:
Participants will be recruited into one of 4 groups according to the Child-Pugh classification score. Participants with HI will be enrolled into either mild (Child-Pugh A; Group 2), moderate (Child Pugh B; Group 3) or severe (Child-Pugh C; Group 4) HI groups. Healthy control participants (Group 1) will be matched to 1 or more participants with HI with respect to age (± 10 years), body weight (± 20%) and sex. Each participant in the matched healthy control group (Group 1) can be matched to participant(s) in any HI group (Groups 2, 3, and 4).

The study will enroll the four groups in parallel. Therefore, enrollment in Group 1 will remain open until enrollment in the mild, moderate and severe HI groups is complete and each HI participant has a matched healthy control (Group 1) participant. Participants from Group 1 will be enrolled after at least 3 participants from each of Groups 2 and 3 have completed all scheduled assessments.

The study consists of a screening period of up to 28 days (Days -29 to -2), a baseline evaluation on Day -1, a single dose administration of siremadlin on Day 1 followed by PK sampling up to 144 hours post-dose (Day 7). All baseline safety evaluation results must be available and reviewed prior to the dosing. All eligible participants will be domiciled from Day -1 until Day 7.

Safety assessments will include physical examinations, ECGs, vital signs, standard clinical laboratory evaluations (hematology, blood chemistry, urinalysis, coagulation), AE and serious adverse event (SAE) monitoring.

All participants will have a post-study safety follow-up contact conducted approximately 30 days after administration of study treatment. The study will be considered complete once all the participants have finished the required assessments, dropped out, or been lost to follow-up before completing the required assessments.

The total study duration for each participant is expected to be up to maximum of 59 days, including the Screening period and the 30-day post-study safety contact follow up period.

ELIGIBILITY:
Key Inclusion Criteria:

All participants:

* Male and non-child-bearing potential females between 18 and 75 years of age, inclusive, at Screening.
* Participant must have been a non-smoker or moderate smoker (up to 10 cigarettes or equivalent nicotine containing products per day) at Screening. Participant must have agreed to maintain the same smoking status (i.e., smoker or non-smoker) from Screening until after Study Completion evaluations.

Additional key inclusion criteria for healthy participants (Group 1):

* Participants must have weighed at least 50.0 kg and must have had a BMI within the range of 18.0 to 38.0 kg/m2, inclusive at Screening.
* Participants with no clinically significant abnormalities as determined by past medical history, physical examination, ECG and clinical laboratory test at Screening.

Additional inclusion criteria for mild, moderate and severe HI participants (Groups 2-4):

* Participants must have weighed at least 50.0 kg and must have had a BMI within the range of 18.0 to 38.0 kg/m2, inclusive at Screening. For participants without overt ascites, the BMI must have been within the range of 18.0 to 40.0 kg/m2, inclusive. For participants with overt ascites, the BMI must have been within the range of 18.0 to 45.0 kg/m2, inclusive.
* Participant must have satisfied the criteria for HI as evidenced by a Child-Pugh class of A, B, or C at Screening and Baseline (see Table 8-2 Child-Pugh classification criteria):

  * Group 2: Class A; Mild; Child-Pugh score 5-6, inclusive
  * Group 3: Class B; Moderate; Child-Pugh score 7-9, inclusive
  * Group 4: Class C; Severe; Child-Pugh score 10-15, inclusive. If the results of the assessments at Screening and Baseline indicated different Child-Pugh class, a third assessment must have been conducted. If the results of the 2 most recent assessments (the second and third) were in agreement with regard to the participant's Child-Pugh class, the participant may have been enrolled at the Child-Pugh class determined by the most recent assessment. If the second and third measurements differ, the participant would not be eligible for the study on the basis that their liver function was not stable.
* Participants with impaired hepatic function and other stable medical disorders such as diabetes, hypertension, hyperlipidemia, hypothyroidism etc., may have been eligible, as long as they were considered appropriate for enrollment, as determined by past medical history, physical examination, vital signs, ECG, and clinical laboratory tests at Screening.

Key Exclusion Criteria:

All participants (Groups 1-4):

* Contraindication or hypersensitivity to the investigational compound/compound class or excipients being used in this study.
* History or presence of clinically significant ECG abnormalities or a family history or presence of prolonged QT-interval syndrome.
* History of malignancy of any organ system, treated or untreated, within 3 years prior to Screening, regardless of whether there were recurrence or metastases. Those with localized basal cell carcinoma of the skin, in-situ cervical cancer, or hepatocellular cancer treated with local ablative therapy more than 6 months prior to Screening may have been enrolled.
* Use of investigational drugs, other than siremadlin (i.e., participation in any clinical investigation) within 4 weeks prior to dosing or longer if required by local regulation, or within 5 half-lives of the investigational agent taken prior to dosing (whichever was longer).
* Clinically significant illness within 2 weeks prior to dosing that may have jeopardized safety of the study participant and/or alter the study results as judged by the Investigator.

Additional key exclusion criteria for healthy participants (Group 1):

* Any single parameter of ALT, AST, GGT, or ALP that exceeded 1.2 x ULN or ≥ 1.5 x ULN TBL or any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or serum TBL at Screening.
* Participants known to have Gilbert's syndrome.
* Participants with abnormal laboratory values for the following parameters at Screening:

  * Hemoglobin levels < 12.0 g/dL (males) or < 11.0 g/dL (females).
  * WBC count outside the range of 3.5 x 109-10.7 x 109 /L (unless deemed not clinically significant by the Investigator).
  * Platelet count < 100 x 109 /L (unless deemed not clinically significant by the Investigator).
* Presence of impaired renal function as indicated by serum creatinine > ULN or abnormal urinary constituents at Screening.

Additional key exclusion criteria for mild and moderate HI participants (Groups 2-3):

* Participants with abnormal laboratory values for the following parameters at Screening:

  * Hemoglobin < 9 g/dL.
  * Platelet count < 30 x 109/L.
  * WBC count < 2.5 x 109/L.
  * TBL > 8 mg/dL.
  * Serum amylase > 5 x ULN with no abdominal symptoms (> 2 x ULN with abdominal symptoms)
  * INR > 2.5.
  * Corrected serum calcium < 8.6 or > 10.2 mg/dL.
* Presence of moderate to severe impaired renal function as indicated by creatinine clearance < 50 mL/min as calculated using the Cockcroft-Gault formula.
* Severe complications of liver disease within the preceding 3 months prior to dosing..
* Trans-jugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.

Additional key exclusion criteria for severe HI participants (Group 4):

* Participants with abnormal laboratory values for the following parameters at Screening:

  * Hemoglobin < 8.5 g/dL.
  * Platelet count < 30 x 109/L.
  * WBC count < 2.5 x 109/L.
  * TBL > 8 mg/dL.
  * Serum amylase > 5 x ULN with no abdominal symptoms (> 2 x ULN with abdominal symptoms).
  * INR > 2.5.
* Presence of moderate to severe impaired renal function as indicated by creatinine clearance < 50 mL/min as calculated using the Cockcroft-Gault formula.
* Severe complications of liver disease within the preceding 3 months prior to dosing.
* Trans-jugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Cmax | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Maximum Observed Blood Concentrations (Cmax) for siremadlin. Blood samples will be collected to measure Cmax at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): AUClast | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Area Under Plasma Concentration-time Curve from time zero to the last measurable concentration sampling time (AUClast) for siremadlin. Blood samples will be collected to measure AUClast at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): AUC0-t | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Area Under Plasma Concentration from time zero to time "t" (AUC0-t). The definition of "t" may be data driven post-hoc to mitigate bias in the exposure comparision due to between-group differences in Tlast for siremadlin. Blood samples will be collected to measure AUC0-t at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): AUC0-24h | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Area Under Plasma Concentration from time zero to 24-hour post-dose sampling time (AUC0-24h) for siremadlin. Blood samples will be collected to measure AUC0-24h at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): Tlast | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Last measurable plasma concentration (Tlast) for siremadlin. Blood samples will be collected to measure Tlast at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): Tmax | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Time to Reach Maximum Blood Concentrations (Tmax) for siremadlin. Blood samples will be collected to measure Tmax at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): CL/F | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Apparent total body clearance of siremadlin from plasma (CL/F). Blood samples will be collected to measure CL/F at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): Vz/F | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Apparent volume of distribution during terminal elimination phase (Vz/F) of siremadlin. Blood samples will be collected to estimate Vz/F at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): T1/2 | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Terminal Elimination Half-life (T1/2) for siremadlin. Blood samples will be collected to measure T1/2 at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.
Pharmacokinetics (PK): AUCinf | pre-dose, 0.5 hours, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, and 144 hours
  Area Under Plasma Concentration from time zero to infinity (AUCinf). Blood samples will be collected to measure AUCinf at indicated timepoints. Pharmacokinetic (PK) parameters will be calculated based on siremadlin blood concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CHDM201X2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18217